CLINICAL TRIAL: NCT01512472
Title: Randomized, Multicentre Efficacy and Safety Study Comparing 10 Mons vs 4 Mons Degarelix Therapy in Prolonging the Off Treatment Interval in Men With Localized Prostate Cancer Receiving Intermittent ADT for Biochemical Recurrence Following Radical Local Therapy
Brief Title: Firmagon (Degarelix) Intermittent Therapy
Acronym: FIT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: acrrual target was not being met
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CURC - FIT-0002
Record Dates: First submitted 2011-11-10; First posted 2012-01-19 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer Recurrent
Keywords: localized prostate cancer; degarelix; intermittent androgen deprivation therapy
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 month degarelix therapy (Active Comparator)
  Interventions: Drug: degarelix
- 4 month degarelix therapy arm (Active Comparator)
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix — Starting dose of 240 mg (40 mg/mL; injection volume 2 x 3 mL; s.c.) degarelix one-month depot will be administered sc on Day 0, followed by a maintenance dose of 80 mg (20 mg/mL; injection volume 1 x 4 mL; s.c.) sc degarelix one-month depot will be administered into the anterior abdominal wall on Month 1, 2, 3, 4, 5, 6, 7, 8 and 9 for the 10 month arm and month 1, 2 and 3 for the 4 month arm.

SUMMARY:
Men with localized prostate cancer requiring intermittent androgen deprivation therapy for biochemical recurrence following radical therapy will be asked to participate in a phase 4 safety and efficacy clinical trial comparing 10 months versus 4 months of degarelix (Firmagon®) therapy with the endpoint of prolonging the off treatment interval.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, randomised trial with subjects receiving subcutaneous (s.c.) monthly injections of degarelix depot. All patients will be treated with a one-month starting dose of 240mg on Day 0. Subjects are then randomized to receive either nine or three maintenance doses of one month duration. The primary objective is to determine the effect of degarelix therapy on the length of the off treatment interval (defined as serum Prostate-specific antigen (PSA) increasing to 5 ng/ml) following completion of the androgen deprivation therapy. The trial will also assess the effect of degarelix therapy on PSA kinetics (specifically PSA doubling time), PSA nadir, and effect on quality of life as well as other measures. The efficacy and safety of these two treatments will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the prostate for which intermittent endocrine treatment therapy is indicated
* PSA level meeting both of these criteria:
* PSA level of ≥ 5 ng/mL.
* For patients with recurrence after radiotherapy or cryotherapy: Patients should have a serum PSA (two measurements) to be >2 ng/mL higher than a previously confirmed PSA nadir.
* screening serum testosterone level above the lower limit of normal range defined as >2.2 ng/mL.

Exclusion Criteria:

* Has had previous or is currently under hormonal management of prostate cancer (surgical castration or other hormonal manipulation)
* Has received therapy with the 5-alpha reductase inhibitors finasteride or dutasteride within 12 weeks and 25 weeks, respectively, prior to screening

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2012-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
serum PSA | approximately 15 months
  The study will compare the length of the off treatment interval (in months) of subjects in the 4 month arm vs those in the 10 month arm. The off treatment interval is defined as the time from PSA nadir following completion of hormone therapy in both arms until the time PSA reaches 5.0ng/ml

SECONDARY OUTCOMES:
serum PSA | at 4 months (4 mon arm) or 10 montths (10 mon arm)
  PSA nadir is described as the serum PSA value after the completion of either 4 months or 10 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — Canadian Urology Research Consortium
Locations (15):
- Canada (15):
  - The Prostate Centre, Vancouver, British Columbia
  - Manitoba Prostate Centre, Winnipeg, Manitoba
  - Centre of Clinical Research, Halifax, Nova Scotia
  - Northeast Cancer Centre, Health Sciences North, Greater Sudbury, Ontario
  - McMaster Institute of Urology, Hamilton, Ontario
  - Centre of Applied Urological Research / Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - URLX Corporation, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Recherches Clinique /Clinical Research, Granby, Quebec
  - The Urology Specialists / Les Urologues Specialises, Montreal, Quebec
  - MUHC Montreal General Hospital, Montreal, Quebec
  - Ultra-Med Research, Pointe-Claire, Quebec
  - Centre de recherche du CHUQ-L'hotel-Dieu de Quebec, Québec, Quebec